CLINICAL TRIAL: NCT02403674
Title: A Phase III Multicenter, Double-Blind, Randomized, Active Comparator-Controlled Clinical Trial to Evaluate the Safety and Efficacy of MK-1439A Once-Daily Versus ATRIPLA™ Once-Daily in Treatment-Naïve HIV-1 Infected Subjects
Brief Title: Comparison of Doravirine, Tenofovir, Lamivudine (MK-1439A) and ATRIPLA™ in Treatment-Naive Human Immunodeficiency Virus Type 1 (HIV-1)-Infected Participants (MK-1439A-021)
Acronym: DRIVE-AHEAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1439A-021; MK-1439A-021 (Other: MSD Protocol Number); 2014-003382-17 (EudraCT Number)
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Human Immunodeficiency Virus (HIV)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — doravirine; Tenofovir; Lamivudine; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doravirine, Tenofovir, Lamivudine (Experimental): Treatment-naive HIV-infected participants will receive doravirine, tenofovir, lamivudine, a single-tablet FDC containing doravirine 100 mg + lamivudine 300 mg + tenofovir disoproxil fumarate 300 mg, q.d. by mouth for 96 weeks. Participants will also take 1 placebo tablet matched to ATRIPLA™ q.d. by mouth for 96 weeks in order to maintain blinding.
  Interventions: Drug: Doravirine, Tenofovir, Lamivudine; Drug: Placebo
- ATRIPLA™ (Active Comparator): Treatment-naive HIV-infected participants will receive ATRIPLA™, a single-tablet FDC containing efavirenz 600 mg + emtricitabine 200 mg + tenofovir disoproxil fumarate 300 mg (equivalent to 245 mg tenofovir disoproxil), q.d. by mouth for 96 weeks. Participants will also take 1 placebo tablet matched to doravirine, tenofovir, lamivudine q.d. by mouth for 96 weeks in order to maintain blinding.
  Interventions: Drug: ATRIPLA™; Drug: Placebo

INTERVENTIONS:
Drug: Doravirine, Tenofovir, Lamivudine — One doravirine, tenofovir, lamivudine tablet taken q.d. by mouth.
  Other Names: MK-1439A
  Arms: Doravirine, Tenofovir, Lamivudine
Drug: ATRIPLA™ — One ATRIPLA™ tablet taken q.d. by mouth
  Arms: ATRIPLA™
Drug: Placebo — Placebo tablets matched to ATRIPLA® or Doravirine, Tenofovir, Lamivudine.

SUMMARY:
The purpose of this study is to compare the antiretroviral activity of doravirine, tenofovir, lamivudine (MK-1439A), a single-tablet, once-daily (q.d.) fixed-dose combination (FDC) containing doravirine (MK-1439A) 100 mg + lamivudine 300 mg + tenofovir disoproxil fumarate 300 mg, with ATRIPLA™, a single-tablet FDC containing efavirenz 600 mg + emtricitabine 200 mg + tenofovir disoproxil fumarate 300 mg, in treatment-naive participants infected with human immunodeficiency virus (HIV). The primary hypothesis is that doravirine, tenofovir, lamivudine q.d. is non-inferior to ATRIPLA™ q.d. as assessed by the proportion of participants with HIV-1 ribonucleic acid (RNA) <50 copies/mL (by the Abbott RealTime HIV-1 Assay) at Week 48. This study has a total duration of 384 weeks, including a 96-week double-blind period and an additional 288-week open-label period.

DETAILED DESCRIPTION:
Participants in Australia, Colombia, Guatemala, Honduras, Israel, New Zealand, Peru, Russia, South Africa, and Thailand who are deriving benefit from doravirine, tenofovir, lamivudine are also eligible to continue receiving study drug during additional open-label extensions which will last for 2 years or until drug is available locally, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Is HIV-1 positive as determined by a positive result on an enzyme-immunoassay, has screening plasma HIV-1 RNA (determined by the central laboratory) ≥1000 copies/mL within 45 days prior to the treatment phase of this study, and has HIV treatment indicated based on physician assessment
* Has never received antiretroviral therapy (ART)
* Is highly unlikely to either become pregnant or impregnate a partner

Exclusion Criteria:

* Has a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound results of the study
* Is a user of recreational or illicit drugs or has a recent history of alcohol/drug abuse
* Has been treated for a viral infection other than HIV-1 (e.g., hepatitis B) with an agent that is active against HIV-1
* Has participated in a study with an investigational drug/device within 30 days prior to Screening
* Has used systemic immunosuppressive therapy or immune modulators within 30 days prior to treatment in this study or is anticipated to need them during the course of the study
* Has a current (active) diagnosis of acute hepatitis due to any cause (note: participants with chronic hepatitis B and C may enter the study as long as they fulfill all entry criteria, have stable liver function tests, and have no significant impairment of hepatic synthetic function)
* Is a female who is pregnant, breastfeeding, or expecting to conceive
* Is a female and is expecting to donate eggs or is male and is expecting to donate sperm (investigators will provide appropriate guidance regarding egg and/or sperm donation after completion of the study treatment regimen)
* Has evidence of decompensated liver disease manifested by the presence of or a history of ascites, esophageal or gastric variceal bleeding, hepatic encephalopathy or other signs or symptoms of advanced liver diseases, or has liver cirrhosis and a Child-Pugh Class C score or Pugh-Turcotte (CPT) score > 9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 734 (Actual)
Dates: Start 2015-06-05 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2023-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Orkin C, Koethe JR, Kumar PN, Sklar P, Xu ZJ, Plank RM, Greaves W, Lahoulou R. Factors Associated With Weight Change After Continuing or Switching to a Doravirine-based Regimen. Open Forum Infect Dis. 2025 Nov 20;12(11):ofaf639. doi: 10.1093/ofid/ofaf639. eCollection 2025 Nov. PMID 41280318
- [Derived] Hsue PY, Behrens GMN, Xu ZJ, Zhao Y, Cmar J, Lahoulou R, Campo RE, Plank RM. Cardiovascular Risk Assessment Using the Atherosclerotic Cardiovascular Disease Risk Score Model after Continuing or Switching to a Doravirine-Based HIV Treatment Regimen. J Acquir Immune Defic Syndr. 2026 Feb 1;101(2):208-213. doi: 10.1097/QAI.0000000000003778. PMID 41081774
- [Derived] Walmsley SL, Kumar PN, Orkin C, Thompson M, Squires K, Xu ZJ, Greaves W, Plank RM, Whiteside Y, Lahoulou R. Efficacy and Safety of Doravirine-based Regimens by Sex and Race: Long-term Results From Three Phase 3 Clinical Trials. Open Forum Infect Dis. 2025 Jul 16;12(7):ofaf356. doi: 10.1093/ofid/ofaf356. eCollection 2025 Jul. PMID 40672760
- [Derived] Moyle G, Meng F, Wan H, Sklar P, Plank RM, Lahoulou R. Brief Report: Resolution of Neuropsychiatric Adverse Events After Switching to a Doravirine-Based Regimen in the Open-Label Extensions of the DRIVE-AHEAD and DRIVE-FORWARD Trials. J Acquir Immune Defic Syndr. 2025 May 1;99(1):81-86. doi: 10.1097/QAI.0000000000003599. PMID 39748155
- [Derived] Orkin C, Molina JM, Cahn P, Lombaard J, Supparatpinyo K, Kumar S, Campbell H, Wan H, Teal V, Jin Xu Z, Asante-Appiah E, Sklar P, Teppler H, Lahoulou R; DRIVE-FORWARD and DRIVE-AHEAD collaborators. Safety and efficacy of doravirine as first-line therapy in adults with HIV-1: week 192 results from the open-label extensions of the DRIVE-FORWARD and DRIVE-AHEAD phase 3 trials. Lancet HIV. 2024 Feb;11(2):e75-e85. doi: 10.1016/S2352-3018(23)00258-8. Epub 2023 Dec 20. PMID 38141637
- [Derived] Orkin C, Squires KE, Molina JM, Sax PE, Sussmann O, Lin G, Kumar S, Hanna GJ, Hwang C, Martin E, Teppler H. Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate (TDF) Versus Efavirenz/Emtricitabine/TDF in Treatment-naive Adults With Human Immunodeficiency Virus Type 1 Infection: Week 96 Results of the Randomized, Double-blind, Phase 3 DRIVE-AHEAD Noninferiority Trial. Clin Infect Dis. 2021 Jul 1;73(1):33-42. doi: 10.1093/cid/ciaa822. PMID 33336698
- [Derived] Orkin C, Molina JM, Lombaard J, DeJesus E, Rodgers A, Kumar S, Martin E, Hanna G, Hwang C. Once-daily Doravirine in Human Immunodeficiency Virus Type 1-Infected, Antiretroviral-naive Adults: An Integrated Efficacy Analysis. Clin Infect Dis. 2020 Mar 17;70(7):1344-1352. doi: 10.1093/cid/ciz424. PMID 31121015
- [Derived] Thompson M, Orkin C, Molina JM, Sax P, Cahn P, Squires K, Xu X, Rodgers A, Kumar S, Teppler H, Martin E, Hanna G, Hwang C. Once-daily Doravirine for Initial Treatment of Adults Living With Human Immunodeficiency Virus-1: An Integrated Safety Analysis. Clin Infect Dis. 2020 Mar 17;70(7):1336-1343. doi: 10.1093/cid/ciz423. PMID 31121013
- [Derived] Orkin C, Squires KE, Molina JM, Sax PE, Wong WW, Sussmann O, Kaplan R, Lupinacci L, Rodgers A, Xu X, Lin G, Kumar S, Sklar P, Nguyen BY, Hanna GJ, Hwang C, Martin EA; DRIVE-AHEAD Study Group. Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate is Non-inferior to Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate in Treatment-naive Adults With Human Immunodeficiency Virus-1 Infection: Week 48 Results of the DRIVE-AHEAD Trial. Clin Infect Dis. 2019 Feb 1;68(4):535-544. doi: 10.1093/cid/ciy540. PMID 30184165
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26049&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment-naïve participants with HIV-1 infection have been recruited at 141 study sites worldwide. The present results include results from the base study (first 96-weeks of the study) along with study extension 1 (week 96-192), study extension 2 (week 192-288), and study extension 3 (week 288-384).
Groups:
- MK-1439A (DOR/3TC/TDF From Day 1): Treatment-naive participants with HIV-1 infection took MK-1439A, a single-tablet fixed dose combination (FDC) containing doravirine (DOR) 100 mg + lamivudine (3TC) 300 mg + tenofovir disoproxil fumarate (TDF) 300 mg, once daily (q.d.) by mouth for 96 weeks. Participants also took 1 placebo tablet matched to ATRIPLA™ q.d. by mouth for 96 weeks in order to maintain blinding. Eligible participants from the Base Study (Day 1 to Week 96) may have entered open-label optional study extensions to receive MK-1439A (FDC containing DOR 100 mg + 3TC 300 mg + TDF 300 mg), taken q.d. during Study Extension 1 (Weeks 96 to 192), Extension 2 (Weeks 192 to 288), and Extension 3 (Weeks 288 to 384).
- ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96): Treatment-naive participants with HIV-1 infection took ATRIPLA™, a single-tablet FDC containing efavirenz (EFV) 600 mg + emtricitabine (FTC) 200 mg + tenofovir disoproxil fumarate (TDF) 300 mg (equivalent to 245 mg tenofovir disoproxil), q.d. by mouth for 96 weeks. Participants also took 1 placebo tablet matched to MK-1439A q.d. by mouth for 96 weeks in order to maintain blinding. Eligible participants from the Base Study (Day 1 to Week 96) may have entered open-label optional study extensions to receive MK-1439A (FDC containing DOR 100 mg + 3TC 300 mg + TDF 300 mg), taken q.d. during Study Extension 1 (Weeks 96 to 192), Extension 2 (Weeks 192 to 288), and Extension 3 (Weeks 288 to 384).
Period: Base Study
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Started (Randomized) | 368 | 366
Treated (Received ≥1 dose of study medication.) | 364 | 364
Completed (Completed through Week 96) | 296 | 276
Not Completed | 72 | 90
Not completed — Death | 1 | 4
Not completed — Adverse Event | 11 | 26
Not completed — Lack of Efficacy | 31 | 23
Not completed — Lost to Follow-up | 6 | 8
Not completed — Withdrawal by Subject | 10 | 17
Not completed — Physician Decision | 2 | 2
Not completed — Pregnancy | 2 | 2
Not completed — Protocol Violation | 8 | 4
Not completed — Non-Compliance with study drug | 1 | 4
Period: Study Extension 1 (Open-Label)
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Started (Not all study participants continued into optional study extension 1) | 291 | 269
Completed | 230 | 205
Not Completed | 61 | 64
Not completed — Adverse Event | 1 | 4
Not completed — Lack of Efficacy | 10 | 13
Not completed — Lost to Follow-up | 8 | 5
Not completed — Withdrawal by Subject | 11 | 13
Not completed — Physician Decision | 2 | 5
Not completed — Pregnancy | 4 | 2
Not completed — Death | 1 | 0
Not completed — Availability of study drug locally | 22 | 19
Not completed — Non-Compliance | 2 | 3
Period: Study Extension 2 (Open-Label)
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Started (Not all study participants continued into optional study extension 2) | 192 | 173
Completed | 150 | 132
Not Completed | 42 | 41
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 1 | 7
Not completed — Withdrawal by Subject | 8 | 6
Not completed — Physician Decision | 1 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Death | 2 | 2
Not completed — Availability of study drug locally | 27 | 23
Not completed — Non-Compliance with study drug | 2 | 0
Period: Study Extension 3 (Open-Label)
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Started (Not all study participants continued into optional study extension 3) | 121 | 111
Completed | 100 | 85
Not Completed | 21 | 26
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Physician Decision | 1 | 5
Not completed — Pregnancy | 0 | 1
Not completed — Availability of study drug locally | 14 | 13

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population consists of all randomized participants who received ≥1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96) | Total
Number analyzed (Participants) | 364 | 364 | 728
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.6 (10.5) | 32.7 (9.9) | 33.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 53 | 112
  Male | 305 | 311 | 616
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 6 | 16
  Asian | 59 | 65 | 124
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 67 | 68 | 135
  White | 177 | 170 | 347
  More than one race | 51 | 55 | 106
  Unknown or Not Reported | 0 | 0 | 0
Baseline cluster of differentiation 4 (CD4) cell counts [Mean (Standard Deviation); unit: cells/mm^3] | 434.9 (217.9) | 415.5 (210.6) | 425.2 (214.3)
Baseline fasting low-density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] — Participants fasted for ≥8 hours prior to LDL-C measurement on Day 1. Population: All randomized participants with baseline data available.
  mg/dL
    number analyzed (Participants) | 353 | 352 | 705
    (all) | 92.08 (32.32) | 90.47 (30.64) | 91.27 (31.48)
Baseline fasting non-high-density lipoprotein cholesterol (non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] — Participants fasted for ≥8 hours prior to non-HDL-C measurement on Day 1. Population: All randomized participants with baseline data available.
  mg/dL
    number analyzed (Participants) | 357 | 357 | 714
    (all) | 115.39 (34.67) | 114.63 (33.55) | 115.01 (34.09)
Baseline fasting cholesterol [Mean (Standard Deviation); unit: mg/dL] — Participants fasted for ≥8 hours prior to cholesterol measurement on Day 1. Population: All randomized participants with baseline data available.
  mg/dL
    number analyzed (Participants) | 357 | 357 | 714
    (all) | 157.29 (36.43) | 156.07 (36.51) | 156.68 (36.45)
Baseline fasting triglycerides [Mean (Standard Deviation); unit: mg/dL] — Participants fasted for ≥8 hour prior to triglycerides measurement on Day 1. Population: All randomized participants with baseline data available.
  mg/dL
    number analyzed (Participants) | 357 | 357 | 714
    (all) | 120.85 (83.06) | 123.23 (82.73) | 122.04 (82.84)
Baseline fasting high-density lipoprotein cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] — Participants fasted for ≥8 hours prior to HDL-C measurement on Day 1. Population: All randomized participants with baseline data available.
  mg/dL
    number analyzed (Participants) | 357 | 357 | 714
    (all) | 41.90 (11.67) | 41.44 (13.08) | 41.67 (12.38)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 Ribonucleic Acid (RNA) <50 Copies/mL at Week 48
Description: The percentage of participants in each arm with HIV-1 RNA levels <50 copies/mL at Week 48 was determined. Plasma HIV-1 RNA levels were quantified with the Abbott RealTime HIV-1 Assay. Data were handled according to the US Food and Drug Administration (FDA) "snapshot" approach in which all missing data are considered treatment failures, regardless of the reason.
Time Frame: Week 48
Population: The analysis population consists of all randomized participants who received ≥1 dose of study medication and had baseline HIV-1 RNA data available.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Number analyzed (Participants) | 364 | 364
Percentage of Participants | 84.3 | 80.8
Statistical Analysis 1: Comparison: MK-1439A (DOR/3TC/TDF From Day 1) vs ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96); Test type: Non-Inferiority — Non-inferiority was declared if the lower bound of the 95% CI of the mean treatment difference was greater than -10; Difference in percentages = 3.537, 95% CI 2-sided [-1.951 to 9.026] — The 95% CIs for difference in percentages were calculated using stratum-adjusted Mantel-Haenszel method for each stratum (HIV-1 RNA ≤100,000 or >100,000 copies/mL)

2. Primary Outcome: Percentage of Participants With Tier-1 Neuropsychiatric Adverse Events (AEs)
Description: The percentage of participants in each arm experiencing ≥1 pre-specified Tier-1 neuropsychiatric AEs was determined. The list of Tier-1 neuropsychiatric AE categories included "dizziness", "sleep disorders and disturbances", and "altered sensorium" (including disturbance in attention).
Time Frame: Up to Week 48
Population: The analysis population consists of all randomized participants who received ≥1 dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Number analyzed (Participants) | 364 | 364
Percentage of Participants
  Dizziness | 8.8 | 37.1
  Sleep disorders and disturbances | 12.1 | 25.5
  Altered sensorium | 4.4 | 8.2
Statistical Analysis 1: Comparison: MK-1439A (DOR/3TC/TDF From Day 1) vs ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96); Dizziness difference; Test type: Superiority — Superiority was declared when the 1-sided p-value comparing treatment difference was <0.02497; p < 0.001, t-test, 2 sided — 2-sided P-value; Difference in percentages = -28.3, 95% CI 2-sided [-34.0 to -22.5] — 95% CIs were calculated using the Miettinen and Nurminen method
Statistical Analysis 2: Comparison: MK-1439A (DOR/3TC/TDF From Day 1) vs ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96); Sleep disorders and disturbances difference; Test type: Superiority — Superiority was declared when the 1-sided p-value comparing treatment difference was <0.02497; p < 0.001, t-test, 2 sided — 2-sided P-value; Difference in percentages = -13.5, 95% CI 2-sided [-19.1 to -7.9] — 95% CIs were calculated using the Miettinen and Nurminen method
Statistical Analysis 3: Comparison: MK-1439A (DOR/3TC/TDF From Day 1) vs ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96); Altered sensorium difference; Test type: Superiority — Superiority was declared when the 1-sided p-value comparing treatment difference was <0.02497; p = 0.033, t-test, 2 sided — 2-sided P-value; Difference in percentages = -3.8, 95% CI 2-sided [-7.6 to -0.3] — 95% CIs were calculated using the Miettinen and Nurminen method

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 96
Description: The percentage of participants in each arm with HIV-1 RNA levels <50 copies/mL at Week 96 were determined. Plasma HIV-1 RNA levels were quantified with the Abbott RealTime HIV-1 Assay. The US Food and Drug Administration (FDA) "snapshot" approach (i.e., all missing data handled as treatment failures, regardless of the reason) were used for efficacy analyses.
Time Frame: Week 96
Population: The analysis population will consist of all randomized participants who received ≥1 dose of study medication and had baseline HIV-1 RNA data available.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Number analyzed (Participants) | 364 | 364
Percentage of participants | 77.5 [72.8 to 81.7] | 73.6 [68.8 to 78.1]
Statistical Analysis 1: Comparison: MK-1439A (DOR/3TC/TDF From Day 1) vs ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96); Test type: Non-Inferiority — Non-inferiority was declared if the lower bound of the 95% CI of the mean treatment difference was greater than -10; Difference in percentages = 3.815, 95% CI 2-sided [-2.412 to 10.042] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA <40 Copies/mL at Week 48
Description: The percentage of participants in each arm with HIV-1 RNA levels <40 copies/mL (including target detected and target not detected) at Week 48 was determined. Plasma HIV RNA levels were quantified with the Abbott RealTime HIV-1 Assay. Data were handled according to the US Food and Drug Administration (FDA) "snapshot" approach in which all missing data are considered treatment failures, regardless of the reason.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Number analyzed (Participants) | 364 | 364
Percentage of Participants | 83.8 [79.6 to 87.4] | 79.7 [75.2 to 83.7]
Statistical Analysis 1: Comparison: MK-1439A (DOR/3TC/TDF From Day 1) vs ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96); Test type: Non-Inferiority — Non-inferiority was declared if the lower bound of the 95% CI of the mean treatment difference was greater than -10; Difference in percentages = 4.1, 95% CI 2-sided [-1.5 to 9.7] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants With HIV-1 RNA <40 Copies/mL at Week 96
Description: The percentage of participants in each arm with HIV-1 RNA levels <40 copies/mL (including target detected and target not detected) at Week 96 were determined. Plasma HIV-1 RNA levels were quantified with the Abbott RealTime HIV-1 Assay. The US Food and Drug Administration (FDA) "snapshot" approach (i.e., all missing data handled as treatment failures, regardless of the reason) were used for efficacy analyses.
Time Frame: Week 96
Population: The analysis population consisted of all randomized participants who received ≥1 dose of study medication and had baseline HIV-1 RNA data available.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Number analyzed (Participants) | 364 | 364
Percentage of participants | 76.1 [71.4 to 80.4] | 72.8 [67.9 to 77.3]
Statistical Analysis 1: Comparison: MK-1439A (DOR/3TC/TDF From Day 1) vs ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96); Test type: Non-Inferiority — Non-inferiority was declared if the lower bound of the 95% CI of the mean treatment difference was greater than -10; Difference in percentages = 3.268, 95% CI 2-sided [-3.057 to 9.593] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change From Baseline in CD4 Cell Counts at Week 48
Description: The mean change from baseline in CD4 cell counts at Week 48 was assessed using the Observed Failure (OF) approach. With the OF approach, baseline values were carried forward for participants who discontinued prior to Week 48 due to lack of efficacy. Cell counts at Baseline and Week 48 were measured and expressed as cells/mm^3, and percent change was then calculated as [(Baseline counts - Week 48 counts)*100]. CD4 cell counts were quantified by a central laboratory using a commercially available assay.
Time Frame: Baseline (Day 1) and Week 48
Population: The analysis population consisted of all randomized participants who received ≥1 dose of study medication and had baseline and Week 48 CD4 data available.
Measure: Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Number analyzed (Participants) | 344 | 329
Percent Change from Baseline | 198.4 [180.2 to 216.7] | 188.4 [169.5 to 207.2]
Statistical Analysis 1: Comparison: MK-1439A (DOR/3TC/TDF From Day 1) vs ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96); Test type: Superiority — Superiority was declared when group difference (MK-1439A-ATRIPLA®) was a positive value; Difference in mean %change from baseline = 10.1, 95% CI 2-sided [-16.1 to 36.3] — 95% CIs were calculated based on t-distribution

7. Secondary Outcome: Change From Baseline in CD4 Cell Counts at Week 96
Description: The mean change from baseline in CD4 cell counts at Week 96 were assessed using the OF approach. With the OF approach, baseline values were carried forward for participants who discontinued prior to Week 96 due to lack of efficacy. Cell counts at Baseline and Week 96 were measured and expressed as cells/mm^3, and percent change was calculated as [(Baseline counts - Week 96 counts)*100]. CD4 cell counts were quantified by a central laboratory using a commercially available assay.
Time Frame: Baseline (Day 1) and Week 96
Population: The analysis population consisted of all randomized participants who received ≥1 dose of study medication and had baseline and week 96 CD4 data available.
Measure: Mean (95% Confidence Interval); unit: Percentage Change from Baseline
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Number analyzed (Participants) | 337 | 311
Percentage Change from Baseline | 237.7 [214.9 to 260.6] | 223.0 [198.4 to 247.6]
Statistical Analysis 1: Comparison: MK-1439A (DOR/3TC/TDF From Day 1) vs ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96); Test type: Superiority — Superiority was declared when group difference (MK-1439A-ATRIPLA) was a positive value; Diff in mean % change from baseline = 14.7, 95% CI 2-sided [-18.7 to 48.2] — The 95% CI for mean difference in CD4 change was based on t-distribution

8. Secondary Outcome: Percentage of Participants Experiencing ≥1 AE
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to Week 48
Population: The analysis population consisted of all randomized participants who received ≥1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Number analyzed (Participants) | 364 | 364
Percentage of participants | 82.7 | 90.7
Statistical Analysis 1: Comparison: MK-1439A (DOR/3TC/TDF From Day 1) vs ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96); Test type: Other — Difference in percentage of participants with ≥1 AE(s); Difference in percentages = -8.0, 95% CI 2-sided [-13.0 to -3.1] — 95% CIs were calculated with the Miettinen & Nurminen method

9. Secondary Outcome: Percentage of Participants Discontinuing From Study Medication Due to an AE(s)
Description: as for outcome 8
Time Frame: Up to Week 48
Population: The analysis population consisted of all randomized participants who received ≥1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Number analyzed (Participants) | 364 | 364
Percentage of participants | 3.0 | 6.6
Statistical Analysis 1: Comparison: MK-1439A (DOR/3TC/TDF From Day 1) vs ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96); Test type: Other — Difference in percentage of participants with ≥1 AE(s); Difference in percentages = -3.6, 95% CI 2-sided [-6.9 to -0.5] — 95% CIs were calculated with the Miettinen & Nurminen method

10. Secondary Outcome: Percentage of Participants With Tier-2 Neuropsychiatric AEs
Description: The percentage of participants in each arm experiencing ≥1 pre-specified Tier-2 neuropsychiatric AEs was determined. The list of Tier-2 neuropsychiatric AE categories included "depression and suicide/self-injury" and "psychosis and psychotic disorders".
Time Frame: Up to Week 48
Population: The analysis population consists of all randomized participants who received ≥1 dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Number analyzed (Participants) | 364 | 364
Percentage of Participants
  Depression and suicide/self-injury | 4.1 | 6.6
  Psychosis and psychotic disorders | 0.3 | 1.1
Statistical Analysis 1: Comparison: MK-1439A (DOR/3TC/TDF From Day 1) vs ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96); Depression and suicide/self-injury difference; Test type: Superiority — Superiority was declared when the 1-sided p-value comparing treatment difference was <0.02497; p < 0.001, t-test, 2 sided — 2-sided P-value; Difference in percentages = -2.5, 95% CI 2-sided [-5.9 to 0.8] — 95% CIs were calculated using the Miettinen and Nurminen method
Statistical Analysis 2: Comparison: MK-1439A (DOR/3TC/TDF From Day 1) vs ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96); Psychosis and psychotic disorders difference; Test type: Superiority — Superiority was declared when the 1-sided p-value comparing treatment difference was <0.02497; p < 0.001, t-test, 2 sided — 2-sided P-value; Difference in percentages = -0.8, 95% CI 2-sided [-2.5 to 0.5] — 95% CIs were calculated using the Miettinen and Nurminen method

11. Secondary Outcome: Change From Baseline in Fasting LDL-C at Week 48
Description: The mean percent change from baseline in fasting (fast duration of ≥8 hours) LDL-C levels at Week 48 was determined for each arm. The Last Observation Carry Forward (LOCF) approach was applied to missing data and data collected after a participant initiated lipid-modifying therapy.
Time Frame: Baseline (Day 1) and Week 48
Population: The analysis population consists of all randomized participants who had baseline LDL-C data available as well as ≥1 LDL-C measurement after initiating study treatment.
Measure: Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Number analyzed (Participants) | 330 | 305
Percent Change from Baseline | -1.58 [-3.98 to 0.81] | 8.74 [5.86 to 11.62]
Statistical Analysis 1: Comparison: MK-1439A (DOR/3TC/TDF From Day 1) vs ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96); Test type: Superiority; p < 0.0001, ANCOVA; Difference in mean %change from baseline = -10.01, 95% CI 2-sided [-13.53 to -6.49] — 95% CIs and 2-sided p-values for treatment difference were calculated from an ANCOVA model with terms for baseline lipid level and treatment

12. Secondary Outcome: Change From Baseline in Fasting Non-HDL-C at Week 48
Description: The mean percent change from baseline in fasting (fast duration of ≥8 hours) non-HDL-C levels at Week 48 was determined for each arm. The LOCF approach was applied to missing data and data collected after a participant initiated lipid-modifying therapy.
Time Frame: Baseline (Day 1) and Week 48
Population: The analysis population consists of all randomized participants who had baseline non-HDL-C data available as well as ≥1 non-HDL-C measurement after initiating study treatment.
Measure: Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Number analyzed (Participants) | 333 | 314
Percent Change from Baseline | -3.83 [-6.27 to -1.40] | 13.26 [10.07 to 16.45]
Statistical Analysis 1: Comparison: MK-1439A (DOR/3TC/TDF From Day 1) vs ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96); Test type: Superiority; p < 0.0001, ANCOVA; Difference in mean %change from baseline = -17.02, 95% CI 2-sided [-20.89 to -13.16] — [estimate comment as in outcome 11, analysis 1]

13. Secondary Outcome: Change From Baseline in Fasting Cholesterol at Week 48
Description: The mean percent change from baseline in fasting (fast duration of ≥8 hours) cholesterol levels at Week 48 was determined for each arm. The LOCF approach was applied to missing data and data collected after a participant initiated lipid-modifying therapy.
Time Frame: Baseline (Day 1) and Week 48
Population: The analysis population consists of all randomized participants who had baseline cholesterol data available as well as ≥1 cholesterol measurement after initiating study treatment.
Measure: Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Number analyzed (Participants) | 333 | 314
Percent Change from Baseline | -1.97 [-4.74 to 0.79] | 21.77 [18.35 to 25.18]
Statistical Analysis 1: Comparison: MK-1439A (DOR/3TC/TDF From Day 1) vs ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96); Test type: Superiority; Difference in mean %change from baseline = -23.44, 95% CI 2-sided [-27.57 to -19.32] — 95% CIs for treatment difference were calculated from an ANCOVA model with terms for baseline lipid level and treatment

14. Secondary Outcome: Change From Baseline in Fasting Triglycerides at Week 48
Description: The mean percent change from baseline in fasting (fast duration of ≥8 hours) triglycerides levels at Week 48 was determined for each arm. The LOCF approach was applied to missing data and data collected after a participant initiated lipid-modifying therapy.
Time Frame: Baseline (Day 1) and Week 48
Population: The analysis population consists of all randomized participants who had baseline triglyceride data available as well as ≥1 triglyceride measurement after initiating study treatment.
Measure: Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Number analyzed (Participants) | 333 | 314
Percent Change from Baseline | -12.40 [-19.66 to -5.15] | 22.01 [11.68 to 32.34]
Statistical Analysis 1: Comparison: MK-1439A (DOR/3TC/TDF From Day 1) vs ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96); Test type: Superiority; Difference in mean %change from baseline = -35.96, 95% CI 2-sided [-47.10 to -24.82] — 95% CIs for treatment difference were calculated from an ANCOVA model with terms for baseline lipid level and treatment

15. Secondary Outcome: Change From Baseline in Fasting HDL-C at Week 48
Description: The mean percent change from baseline in fasting (fast duration of ≥8 hours) HDL-C levels at Week 48 was determined for each arm. The LOCF approach was applied to missing data and data collected after a participant initiated lipid-modifying therapy.
Time Frame: Baseline (Day 1) and Week 48
Population: The analysis population consists of all randomized participants who had baseline HDL-C data available as well as ≥1 HDL-C measurement after initiating study treatment.
Measure: Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Number analyzed (Participants) | 333 | 314
Percent Change from Baseline | 1.86 [0.83 to 2.89] | 8.51 [7.32 to 9.69]
Statistical Analysis 1: Comparison: MK-1439A (DOR/3TC/TDF From Day 1) vs ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96); Test type: Superiority; Difference in mean %change from baseline = -6.47, 95% CI 2-sided [-7.97 to -4.96] — 95% CIs for treatment difference were calculated from an ANCOVA model with terms for baseline lipid level and treatment

16. Secondary Outcome: Percentage of Participants With HIV-1 RNA Below the Limit of Quantification (BLoQ) at Week 48
Description: The percentage of participants in each arm with HIV-1 RNA levels BLoQ of 40 copies/mL and target not detected at Week 48 was determined. Plasma HIV RNA levels were quantified with the Abbott RealTime HIV-1 Assay. Data were handled as observed.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Number analyzed (Participants) | 364 | 364
Percentage of Participants | 59.6 | 55.5

17. Secondary Outcome: Percentage of Participants With HIV-1 RNA BLoQ at Week 96
Description: The percentage of participants in each arm with HIV-1 RNA levels BLoQ of 40 copies/mL and target not detected at Week 96 was determined. Plasma HIV RNA levels was quantified with the Abbott RealTime HIV-1 Assay. Data was handled as observed.
Time Frame: Week 96
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1) | ATRIPLA™ (Switch From EFV/FTC/TDF at Week 96)
Number analyzed (Participants) | 364 | 364
Percentage of Participants | 59.3 | 59.1

18. Secondary Outcome: Plasma Concentration of Doravirine at Week 48
Description: Plasma samples were collected for analysis of doravirine concentration at Week 48. A total of 2 samples were collected: 1 prior to dosing and 1 collected between 0.5 and 2 hours post-dose.
Time Frame: 0 hours post-dose and 2 hours post-dose on Week 48
Population: The analysis population consists of all randomized participants in the MK-1439A arm who received ≥1 dose of study drug and had doravirine concentration data available.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | MK-1439A (DOR/3TC/TDF From Day 1)
Number analyzed (Participants) | 312
nM
  Pre-dose | 1290 (799)
  0.5 to 2 hours post-dose: number analyzed (Participants) | 310
  0.5 to 2 hours post-dose | 2330 (1230)

ADVERSE EVENTS:
Time Frame: Up to 430 weeks
Description: All cause-mortality was reported on all allocated participants. Serious and non-serious AEs were reported for all allocated participants who received ≥1 dose of study treatment. Per protocol, serious adverse events and all-cause mortality were collected up to 430 weeks, and non-serious adverse event data were collected up to 192 weeks.
Groups:
- DOR/3TC/TDF Only (From Day 1) at Base Study: Treatment-naive participants took a single-tablet FDC containing doravirine 100 mg + lamivudine 300 mg + tenofovir disoproxil fumarate 300 mg, q.d. by mouth for a total of 96 weeks.
- DOR/3TC/TDF Switch at Week 96 Base Study: Treatment-naive participants with HIV-1 infection took ATRIPLA™, a single-tablet FDC containing efavirenz 600 mg + emtricitabine 200 mg + tenofovir disoproxil fumarate 300 mg (equivalent to 245 mg tenofovir disoproxil), q.d. by mouth for a total of 96 weeks.
- DOR/3TC/TDF Only (DOR/3TC/TDF From Day 1) Ext 1; DOR/3TC/TDF Switch (Switch From EFV/FTC/TDF at Week 96) Ext 1: One doravirine, tenofovir, lamivudine taken q.d. by mouth for an additional 96 weeks (Week 96 - Week 192)
- DOR/3TC/TDF Only (DOR/3TC/TDF From Day 1) Ext 2; DOR/3TC/TDF Switch (Switch From EFV/FTC/TDF at Week 96) Ext 2: One doravirine, tenofovir, lamivudine taken q.d. by mouth for an additional 96 weeks (Week 192 - Week 288)
- DOR/3TC/TDF Only (DOR/3TC/TDF From Day 1) Ext 3; DOR/3TC/TDF Switch (Switch From EFV/FTC/TDF at Week 96) Ext 3: One doravirine, tenofovir, lamivudine taken q.d. by mouth for an additional 96 weeks (Week 388 - Week 384)
Arm/Group | DOR/3TC/TDF Only (From Day 1) at Base Study | DOR/3TC/TDF Switch at Week 96 Base Study | DOR/3TC/TDF Only (DOR/3TC/TDF From Day 1) Ext 1 | DOR/3TC/TDF Switch (Switch From EFV/FTC/TDF at Week 96) Ext 1 | DOR/3TC/TDF Only (DOR/3TC/TDF From Day 1) Ext 2 | DOR/3TC/TDF Switch (Switch From EFV/FTC/TDF at Week 96) Ext 2 | DOR/3TC/TDF Only (DOR/3TC/TDF From Day 1) Ext 3 | DOR/3TC/TDF Switch (Switch From EFV/FTC/TDF at Week 96) Ext 3
All-Cause Mortality (participants affected / at risk) | 1/368 | 4/366 | 2/291 | 0/269 | 2/192 | 2/173 | 0/121 | 0/111
Serious Adverse Events (participants affected / at risk) | 22/364 | 30/364 | 19/291 | 12/269 | 8/192 | 9/173 | 2/121 | 7/111
Other Adverse Events (participants affected / at risk) | 231/364 | 281/364 | 111/291 | 110/269 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOR/3TC/TDF Only (From Day 1) at Base Study (N=364) | DOR/3TC/TDF Switch at Week 96 Base Study (N=364) | DOR/3TC/TDF Only (DOR/3TC/TDF From Day 1) Ext 1 (N=291) | DOR/3TC/TDF Switch (Switch From EFV/FTC/TDF at Week 96) Ext 1 (N=269) | DOR/3TC/TDF Only (DOR/3TC/TDF From Day 1) Ext 2 (N=192) | DOR/3TC/TDF Switch (Switch From EFV/FTC/TDF at Week 96) Ext 2 (N=173) | DOR/3TC/TDF Only (DOR/3TC/TDF From Day 1) Ext 3 (N=121) | DOR/3TC/TDF Switch (Switch From EFV/FTC/TDF at Week 96) Ext 3 (N=111)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid cyst (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis A (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oophoritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pilonidal disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic nodular goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orchitis mumps (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurosyphilis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myopericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaplastic large-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mania (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOR/3TC/TDF Only (From Day 1) at Base Study (N=364) | DOR/3TC/TDF Switch at Week 96 Base Study (N=364) | DOR/3TC/TDF Only (DOR/3TC/TDF From Day 1) Ext 1 (N=291) | DOR/3TC/TDF Switch (Switch From EFV/FTC/TDF at Week 96) Ext 1 (N=269) | DOR/3TC/TDF Only (DOR/3TC/TDF From Day 1) Ext 2 (N=0) | DOR/3TC/TDF Switch (Switch From EFV/FTC/TDF at Week 96) Ext 2 (N=0) | DOR/3TC/TDF Only (DOR/3TC/TDF From Day 1) Ext 3 (N=0) | DOR/3TC/TDF Switch (Switch From EFV/FTC/TDF at Week 96) Ext 3 (N=0)
Diarrhoea (Gastrointestinal disorders) | 50 (73) | 58 (68) | 16 (21) | 17 (18) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 31 (35) | 42 (55) | 5 (5) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 19 (23) | 29 (42) | 1 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 22 (25) | 24 (26) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 50 (89) | 43 (61) | 40 (58) | 26 (36) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 30 (39) | 20 (27) | 13 (16) | 11 (18) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 41 (55) | 30 (40) | 21 (33) | 19 (22) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (23) | 19 (21) | 7 (7) | 14 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 37 (47) | 139 (155) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 58 (96) | 56 (77) | 18 (19) | 16 (21) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 13 (13) | 28 (28) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 18 (20) | 44 (49) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 24 (35) | 38 (42) | 6 (7) | 10 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (25) | 20 (24) | 8 (8) | 11 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 20 (22) | 50 (54) | 8 (9) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syphilis (Infections and infestations) | 18 (21) | 14 (15) | 16 (18) | 15 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT02403674/Prot_SAP_001.pdf